CLINICAL TRIAL: NCT00586911
Title: A Randomized, Placebo-Controlled Trial of Betaine in Patients With Nonalcoholic Steatohepatitis (NASH)
Brief Title: Betaine in Patients With Nonalcoholic Steatohepatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of Florida (Other); Orphan Medical (Industry)
Responsible Party: Dr. Keith D. Lindor, MD / PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 458-00
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: Nonalcoholic Steatohepatitis; NASH; Betaine
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Betaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cystadane (Active Comparator)
  Interventions: Drug: Cystadane
- Identical Placebo (Placebo Comparator)
  Interventions: Drug: Identical Placebo

INTERVENTIONS:
Drug: Cystadane — Betaine 20 mg a day or identical placebo for 1 year.
  Arms: Cystadane
Drug: Identical Placebo — Placebo
  Arms: Identical Placebo

SUMMARY:
To assess the safety and efficacy of betaine in patients with NASH on markers of disease severity such as liver histology, liver biochemistries, and health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females, age 18 - 70 (inclusive) with NASH.
* Abnormal aminotransferase levels (1.5x normal) on at least two occasions at less three months apart.
* Histologic evidence of steatohepatitis on liver biopsy performed within six months of entry.
* Absence of sustained alcohol ingestion (less than 20 g/d in women or 30 g/d in men).
* Compensated liver disease and blood cell counts within the following limits: Hb > 12 gr/dl, platelets > 120,000/mm3, and WBC > 3,000/mm3
* TSH (thyroid-stimulating hormone) within normal limits of testing laboratory.
* Appropriate exclusion of other liver disease such as viral, autoimmune and metabolic/hereditary liver disease.
* If a history of diabetes, a hemoglobin A1C < 10.0%.
* Alpha-fetoprotein in normal range (obtained within the previous year), or if greater than normal, the patient requires a negative ultrasound for hepatocellular carcinoma within prior 3 months.
* Sexually active female patients of childbearing potential must practice adequate contraception during the treatment period and for 6 months after discontinuation of therapy. A pregnancy test obtained at entry prior to the initiation of treatment must by negative. Female patients must not be breast-feeding.
* Sexually active male patients must practice acceptable methods of contraception during the treatment period and for 6 months after discontinuation of therapy.
* Written informed consent for participation in this study.

Exclusion Criteria:

* Treatment with any experimental drug for NASH, betaine, ursodeoxycholic acid (URSO), methionine, rosiglitazone, metformin, pioglitazone, or vitamin E within 3 months of enrollment or at time of pre-entry liver biopsy. (Patients with diabetes and on stable medical management for six months prior to entry and an anticipated stable program throughout the study will be eligible. Medications that may be used include insulin, biguanides, thiazolidnediones, metformin, and sulfonylureas. Patients with hyperlipidemia on a medical program for control of lipids who have had a change in drug treatment in the preceding six months or with anticipated changes in the year of the study will also be eligible.)
* Any cause for the liver disease based on patient history and biopsy (where applicable) other than NASH
* Evidence of decompensated liver disease such as history or presence of ascites, bleeding varices, spontaneous encephalopathy.
* Any known pre-existing medical condition that could interfere with the patient's participation in and completion of the study such as significant cardiovascular dysfunction or chronic obstructive pulmonary disease requiring specific therapy
* Pregnancy or breastfeeding.
* Unwillingness of patient and/or partner to use contraception during treatment.
* Previous malignant disease (other than non-melanoma skin cancer) in the previous two years.
* Substance abuse, such as alcohol, I.V. drugs and inhaled drugs.
* Any other conditions that in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in and completing the protocol.
* Lactose intolerant patient since placebo preparation contains lactose.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2003-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
changes in degree of steatosis, necroinflammatory activity and fibrosis in liver biopsy. | 1 year

SECONDARY OUTCOMES:
Secondary end-points will be changes in liver test results and health related quality of life. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Keith D Lindor, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - University of Florida at Gainesville, Gainesville, Florida
  - Mayo Clinic, Rochester, Minnesota